CLINICAL TRIAL: NCT05329610
Title: β-alanine Supplementation in Adults With Overweight or Obesity (BASA-O): A Randomised Controlled Feasibility Trial
Brief Title: β-alanine Supplementation in Adults With Overweight/Obesity
Acronym: BASA-O
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nottingham Trent University (Other)
Collaborators: Aston University (Other)
Responsible Party: Principal Investigator, Joseph J Matthews, PhD Researcher, Nottingham Trent University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 676
Record Dates: First submitted 2021-10-21; First posted 2022-04-15 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Prediabetes; Hyperglycemia; Overweight or Obesity
Keywords: Prediabetes; Hyperglycemia; Carnosine; Overweight; Obesity
MeSH Terms: conditions — Prediabetic State; Hyperglycemia; Overweight; Obesity | interventions — beta-Alanine

STUDY DESIGN:
Intervention Model Description: A double-blinded, randomised, placebo-controlled, parallel group, feasibility trial. The allocation ratio of treatment to placebo will be 1:1.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: All participants, data collectors, and outcome assessors will be blind to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beta-alanine (Experimental): Slow-release beta-alanine (Natural Alternatives International, Carlsbad, CA, USA). Dose: 4.8 grams per day for 3-months (potential total intake of 432 g beta-alanine). The daily intake will be split into four doses of 2 x 600 mg. Participants will be instructed to consume each dose alongside their main daily meals (e.g., breakfast, lunch, and dinner) and before bed.
  Interventions: Dietary Supplement: Beta-alanine
- Placebo (Placebo Comparator): Taste and appearance-matched placebo (tapioca starch) (Natural Alternatives International, Carlsbad, CA, USA). Doses equivalent to the experimental arm.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Beta-alanine — Slow-release beta-alanine.
  Arms: Beta-alanine
Dietary Supplement: Placebo — Taste and appearance-matched placebo (tapioca starch).
  Arms: Placebo

SUMMARY:
The study will investigate the safety, feasibility, and efficacy of beta-alanine supplementation in adults with overweight or obesity. Beta-alanine is a widely used dietary supplement that can increase the amount of carnosine in skeletal muscle. Both carnosine and beta-alanine occur naturally in animal food products and previous research shows that supplementation with beta-alanine leads to an improvement in exercise performance; more recently, the present investigators have shown that increasing carnosine can also help to improve cardiometabolic health, detoxify skeletal muscle, and improve glucose (sugar) uptake into muscle cells.

The investigators will recruit 30 participants (15 per arm) with overweight or obesity who meet the study criteria (this accounts for up to 20% attrition - a minimum of 12 participants per arm). Those who are eligible will be required to receive three short telephone calls and attend three laboratory sessions. Participants will be randomised to receive either beta-alanine or placebo (an inactive sugar pill) for the 3-month study period.

To see whether beta-alanine supplementation is feasible in this population the investigators will measure recruitment, adherence (how well people can stick to the supplement regime), the number and nature of side effects, and blinding to the intervention. Markers of cardiac function, glycaemic control, and metabolic health will also be explored. All measurements will take place before and after a 3-month supplementation period. This will provide us with novel information of the role of beta-alanine and carnosine in cardiometabolic health; and will aid in the planning of a larger randomised controlled trial to assess the efficacy of beta-alanine supplementation as a therapeutic strategy.

DETAILED DESCRIPTION:
Overweight and obesity are major public health problems. Recent estimates show that 64.3% of people in the UK are living with overweight or obesity; this is projected to increase to 71% by 2040, which equates to approx. 42.2 million people (Cancer Research UK, 2022). Overweight and obesity are characterised by excess amounts of adiposity and systemic, chronic, low-grade inflammation, which is associated with a range of metabolic disorders including dyslipidaemia, hypertension, and hyperglycaemia (Calder et al., 2011). This confers an increased risk of developing prediabetes, type-2 diabetes, and cardiovascular disease, as well as associated microvascular complications such as retinopathy, neuropathy, and nephropathy (Brannick et al., 2016). Lifestyle interventions can help delay or prevent the progression of overweight or obesity, thereby reducing morbidity (Lin et al., 2017; Wing et al., 2021). Such interventions, however, can be challenging to implement and a lack of long-term adherence can limit their effectiveness (Fappa et al., 2008). It is therefore important to develop low-cost, novel adjunct therapies to improve cardiometabolic health and help delay or prevent disease progression.

The multifunctional dipeptide carnosine has emerged as a candidate for improving glycaemic control and cardiometabolic health. A recent meta-analysis showed that supplementation with carnosine, or its rate-limiting precursor β-alanine, reduces fasting glucose and HbA1c in humans and rodents. Work from our Research Group shows that treatment with carnosine decreases highly toxic lipid peroxidation products in skeletal muscle cells, leading to an increase in insulin-stimulated glucose uptake under glucolipotoxic conditions. A similar role occurs in vivo, where supplementation with β-alanine leads to greater formation of carnosine-adducts in post-exercise skeletal muscle samples. Given that skeletal muscle insulin resistance is a key component of prediabetes and type 2 diabetes, and reactive aldehydes can directly interfere with insulin signalling, carnosine may exert its therapeutic actions in skeletal muscle. There is also emerging evidence that carnosine, and other histidine-containing dipeptides (HCDs), play an important role in Ca2+ handling and excitation-contraction coupling in cardiac muscle, which may have implications for cardiovascular health. A limitation of existing studies is that the low carnosine dose used is likely to have only a modest effect on tissue carnosine content. Supplementation with β-alanine, however, can increase skeletal muscle carnosine content by 60-80% in 4-10 weeks, but it has not yet been trialled in adults with overweight or obesity.

Please note: a change was made to the study eligibility criteria, which was approved by the UK Health Research Authority Research Ethics Committee on 01/09/2022.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 to 75 years
* Body Mass Index (BMI) ≥25 to <40 kg/m2
* Able to provide informed consent

Exclusion Criteria:

* Weight loss or gain ≥5 kg in the prior 6 months
* Current participation in another clinical research trial
* Substance abuse, presence of an eating disorder or purging behaviour
* Known mental health illness requiring active treatment
* Known cognitive impairment
* Inability to understand conversational English
* Presence of type-1 or type-2 diabetes mellitus
* Use of carnosine or β-alanine supplements in the prior 6 months
* Current breastfeeding, pregnancy, or consideration of pregnancy
* Known comorbidities which may impact on study aims (e.g., cancer, heart failure, or chronic kidney disease) or measurement of study outcomes (e.g., sickle cell anaemia or previously known haemoglobinopathy)
* Use of weight loss or glucose lowering drugs (e.g., orlistat, thyroxine, metformin, insulin, glucagon-like-peptide-1 analogues), long-term corticosteroids, or other drugs which may impact on measurement of study outcomes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Adherence to the intervention | 3-months (endpoint)
  Probability that a randomised participant receives the assigned intervention.

SECONDARY OUTCOMES:
Recruitment | Baseline
  Probability an eligible participant consents and is randomised.
Attrition rate | 3-months (endpoint)
  Probability that a randomised participant is evaluated for baseline and follow-up.
Side effects | Baseline and 3-months (endpoint)
  Data collected using the GASE questionnaire.
Blinding to the intervention | 3-months (endpoint)
  Assessed using the -1, 0, +1 scale (Bang et al., 2004).

OTHER OUTCOMES:
Body weight (kg) | Baseline and 3-months (endpoint)
  Body weight will be measured with minimal clothing, using calibrated scales, and recorded to the nearest 0.1 kg.
BMI (kg/m2) | Baseline and 3-months (endpoint)
  Body mass index will be calculated from these measures, using the standard formula: [weight (kg) / height2 (m)].
Waist circumference (cm) | Baseline and 3-months (endpoint)
  Waist circumference will be taken as the circumference of the abdomen at its narrowest point, between the lower costal border and the top of the iliac crest.
Hand grip strength (kg) | Baseline and 3-months (endpoint)
  Hand grip strength will be measured using the standardised Southampton grip-strength protocol (Roberts et al., 2011).
HbA1c (glycated haemoglobin) | Baseline and 3-months (endpoint)
  Analyses will be performed using a Quo-Lab® HbA1c Analyzer (EKF Diagnostics, Germany).
Fasting plasma glucose | Baseline and 3-months (endpoint)
  Analyses will be performed using a Clinical Chemistry Analyser (ABX Pentra C400, Bergman Diagnostica, Horiba Medical, France).
Fasting plasma insulin | Baseline and 3-months (endpoint)
  Analyses will be performed using commercially available kits (e.g., enzyme-linked immunosorbent assays) and other relevant analytical methods.
Plasma C-peptide | Baseline and 3-months (endpoint)
  Analyses will be performed using commercially available kits (e.g., enzyme-linked immunosorbent assays) and other relevant analytical methods.
Homeostatic model assessment of insulin sensitivity (HOMA2-S%) | Baseline and 3-months (endpoint)
  HOMA2-S% will be used to estimate insulin sensitivity using the Oxford computer method (available from https://dtu.ox.ac.uk/homacalculator/) (Wallace et al., 2004).
Homeostatic model assessment of beta-cell function (HOMA2-β%) | Baseline and 3-months (endpoint)
  HOMA2-β% will be used to estimate β-cell function using the Oxford computer method (available from https://dtu.ox.ac.uk/homacalculator/) (Wallace et al., 2004).
Quantitative insulin sensitivity check index (QUICKI) | Baseline and 3-months (endpoint)
  The QUICKI will be used as an additional measure of insulin sensitivity, using the standard formula: QUICKI = 1 / [log(fasting insulin) + log(fasting glucose)] (Katz et al., 2000).
Plasma fructosamine | Baseline and 3-months (endpoint)
  Analyses will be performed using a Clinical Chemistry Analyser (ABX Pentra C400, Bergman Diagnostica, Horiba Medical, France).
Plasma C-reactive protein | Baseline and 3-months (endpoint)
  Analyses will be performed using a Clinical Chemistry Analyser (ABX Pentra C400, Bergman Diagnostica, Horiba Medical, France).
Plasma lipids and profile | Baseline and 3-months (endpoint)
  High density lipoprotein (HDL), low density lipoprotein (LDL), total cholesterol (TC), triglycerides, LDL:HDL, and TC:HDL. Analyses will be performed using a Clinical Chemistry Analyser (ABX Pentra C400, Bergman Diagnostica, Horiba Medical, France).
Plasma apolipoprotein A-1 | Baseline and 3-months (endpoint)
  Analyses will be performed using a Clinical Chemistry Analyser (ABX Pentra C400, Bergman Diagnostica, Horiba Medical, France), commercially available kits (e.g., enzyme-linked immunosorbent assays) and other relevant analytical methods.
Plasma apolipoprotein B | Baseline and 3-months (endpoint)
  Analyses will be performed using a Clinical Chemistry Analyser (ABX Pentra C400, Bergman Diagnostica, Horiba Medical, France), commercially available kits (e.g., enzyme-linked immunosorbent assays) and other relevant analytical methods.
Plasma and urine markers of carnosine and carnosinase metabolism | Baseline and 3-months (endpoint)
  Blood and urine analyses will be performed using commercially available kits (e.g., enzyme-linked immunosorbent assays) and other relevant analytical methods.
Plasma and urine markers of oxidative stress, glycation, and lipid peroxidation | Baseline and 3-months (endpoint)
  Blood and urine analyses will be performed using commercially available kits (e.g., enzyme-linked immunosorbent assays) and other relevant analytical methods.
Liver function: alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase, gamma-glutamyl transferase, lactate dehydrogenase, creatine kinase (U/L). | Baseline and 3-months (endpoint)
  Blood analyses will be performed using a Clinical Chemistry Analyser (ABX Pentra C400, Bergman Diagnostica, Horiba Medical, France); commercially available kits (e.g., enzyme-linked immunosorbent assays); and other relevant analytical methods.
Liver function: albumin and total protein (g/L) | Baseline and 3-months (endpoint)
  Blood analyses will be performed using a Clinical Chemistry Analyser (ABX Pentra C400, Bergman Diagnostica, Horiba Medical, France); commercially available kits (e.g., enzyme-linked immunosorbent assays); and other relevant analytical methods.
Kidney and liver function: serum creatinine and total bilirubin (µmol/L) | Baseline and 3-months (endpoint)
  Blood analyses will be performed using a Clinical Chemistry Analyser (ABX Pentra C400, Bergman Diagnostica, Horiba Medical, France); commercially available kits (e.g., enzyme-linked immunosorbent assays); and other relevant analytical methods.
Kidney function: urea (mmol/L) | Baseline and 3-months (endpoint)
  Blood analyses will be performed using a Clinical Chemistry Analyser (ABX Pentra C400, Bergman Diagnostica, Horiba Medical, France); commercially available kits (e.g., enzyme-linked immunosorbent assays); and other relevant analytical methods.
Estimated glomerular filtration rate (eGFR) (mL/min/1.73m2). | Baseline and 3-months (endpoint)
  Calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation, which uses serum creatinine (µmol/L), age, sex, and race.
Urinary albumin:creatinine ratio (mg/mmol) | Baseline and 3-months (endpoint)
  Calculated from measurements of urine albumin (mg/L) and urine creatinine (µmol/L).
N-terminal pro-brain natriuretic peptide (NT-proBNP) | Baseline and 3-months (endpoint)
  Analyses will be performed using commercially available kits (e.g., enzyme-linked immunosorbent assays) and other relevant analytical methods.
Diastolic, systolic, and meal arterial blood pressures (mmHg) | Baseline and 3-months (endpoint)
  Non-invasive continuous haemodynamic measurements will be recorded using the CNAP Monitor (CNSystems, Graz; Austria), which uses fingertip plethysmography to accurately measure the beat-to-beat blood pressure wave form; or SBP/DBP will be measured using an automated sphygmomanometer.
Cardiac output (L/min) | Baseline and 3-months (endpoint)
  Calculated from measurements of stroke volume (mL) and heart rate (bpm), using the CNAP Monitor (CNSystems, Graz; Austria); and/or from resting transthoracic echocardiographic (TTE) measurements using a portable ultrasound system (Siemens, USA) and a 4 mHz cardiac transducer.
Stroke volume index (mL/m2) | Baseline and 3-months (endpoint)
  Calculated using body index from measurements using the CNAP Monitor (CNSystems, Graz; Austria); and/or from resting transthoracic echocardiographic (TTE) measurements using a portable ultrasound system (Siemens, USA) and a 4 mHz cardiac transducer.
Cardiac index (L/min/m2) | Baseline and 3-months (endpoint)
  Calculated using body index from measurements using the CNAP Monitor (CNSystems, Graz; Austria); and/or from resting transthoracic echocardiographic (TTE) measurements using a portable ultrasound system (Siemens, USA) and a 4 mHz cardiac transducer.
Systemic vascular resistance (SVR) (dyne*s/cm5) | Baseline and 3-months (endpoint)
  Calculated using cardiac output (L/min) and mean arterial pressure (mmHg).
Systemic vascular resistance (SVR) (dyne*s*m2/cm5) | Baseline and 3-months (endpoint)
  Calculated using cardiac output (L/min), mean arterial pressure (mmHg), and body index.
Isovolumetric contraction and relaxation times (IVCT/IVRT) (ms) | Baseline and 3-months (endpoint)
  Calculated from resting transthoracic echocardiographic (TTE) measurements using a portable ultrasound system (Siemens, USA) and a 4 mHz cardiac transducer.
Left ventricular ejection fraction and systolic function (LVEF/LVSF) (%) | Baseline and 3-months (endpoint)
  Calculated from resting transthoracic echocardiographic (TTE) measurements using a portable ultrasound system (Siemens, USA) and a 4 mHz cardiac transducer.
End systolic and diastolic volumes (mL) | Baseline and 3-months (endpoint)
  Calculated from resting transthoracic echocardiographic (TTE) measurements using a portable ultrasound system (Siemens, USA) and a 4 mHz cardiac transducer.
Left ventricle systolic and diastolic diameters (mm) | Baseline and 3-months (endpoint)
  Calculated from resting transthoracic echocardiographic (TTE) measurements using a portable ultrasound system (Siemens, USA) and a 4 mHz cardiac transducer.
Myocardial performance index (MPI) (also known as Tei Index; TI) | Baseline and 3-months (endpoint)
  Calculated from the sum of isovolumic contraction time (ICT) and isovolumic relaxation time (IRT) divided by ejection time (ET).
Ejection time (ms) | Baseline and 3-months (endpoint)
  Calculated from resting transthoracic echocardiographic (TTE) measurements using a portable ultrasound system (Siemens, USA) and a 4 mHz cardiac transducer.
Aortic blood flow and A-Vmax (cm/s) | Baseline and 3-months (endpoint)
  Calculated from resting transthoracic echocardiographic (TTE) measurements using a portable ultrasound system (Siemens, USA) and a 4 mHz cardiac transducer.
E wave deceleration time (DT) (ms) | Baseline and 3-months (endpoint)
  Calculated from resting transthoracic echocardiographic (TTE) measurements using a portable ultrasound system (Siemens, USA) and a 4 mHz cardiac transducer.
E wave (m/s) | Baseline and 3-months (endpoint)
  Calculated from resting transthoracic echocardiographic (TTE) measurements using a portable ultrasound system (Siemens, USA) and a 4 mHz cardiac transducer.
A wave (m/s) | Baseline and 3-months (endpoint)
  Calculated from resting transthoracic echocardiographic (TTE) measurements using a portable ultrasound system (Siemens, USA) and a 4 mHz cardiac transducer.
E/A ratio | Baseline and 3-months (endpoint)
  Calculated from resting transthoracic echocardiographic (TTE) measurements using a portable ultrasound system (Siemens, USA) and a 4 mHz cardiac transducer.
E' | Baseline and 3-months (endpoint)
  Calculated from resting transthoracic echocardiographic (TTE) measurements using a portable ultrasound system (Siemens, USA) and a 4 mHz cardiac transducer.
e/e' | Baseline and 3-months (endpoint)
  Calculated from resting transthoracic echocardiographic (TTE) measurements using a portable ultrasound system (Siemens, USA) and a 4 mHz cardiac transducer.
Left and right ventricular dimensions (mm) | Baseline and 3-months (endpoint)
  Calculated from resting transthoracic echocardiographic (TTE) measurements using a portable ultrasound system (Siemens, USA) and a 4 mHz cardiac transducer.
Left and right ventricular areas and atrial area (cm/2) | Baseline and 3-months (endpoint)
  Calculated from resting transthoracic echocardiographic (TTE) measurements using a portable ultrasound system (Siemens, USA) and a 4 mHz cardiac transducer.
Left and right ventricular outflow tract views (LVOT/RVOT) (mm or cm) | Baseline and 3-months (endpoint)
  Calculated from resting transthoracic echocardiographic (TTE) measurements using a portable ultrasound system (Siemens, USA) and a 4 mHz cardiac transducer.
Left and right diastolic function (cm/s) | Baseline and 3-months (endpoint)
  Calculated from resting transthoracic echocardiographic (TTE) measurements using a portable ultrasound system (Siemens, USA) and a 4 mHz cardiac transducer.
Right ventricular fractional area change (RVFAC) (%) | Baseline and 3-months (endpoint)
  Calculated from resting transthoracic echocardiographic (TTE) measurements using a portable ultrasound system (Siemens, USA) and a 4 mHz cardiac transducer.
Left and right ventricle tissue doppler imaging (LVTDI/RVTDI) (cm/s) | Baseline and 3-months (endpoint)
  Calculated from resting transthoracic echocardiographic (TTE) measurements using a portable ultrasound system (Siemens, USA) and a 4 mHz cardiac transducer.
Left ventricle longitudinal, circumferential, and radial strain | Baseline and 3-months (endpoint)
  Calculated from resting transthoracic echocardiographic (TTE) measurements using a portable ultrasound system (Siemens, USA) and a 4 mHz cardiac transducer. Reported as % or % per second.
Left ventricle twist and untwist mechanics | Baseline and 3-months (endpoint)
  Calculated from resting transthoracic echocardiographic (TTE) measurements using a portable ultrasound system (Siemens, USA) and a 4 mHz cardiac transducer. Reported as degrees or degrees per second.
Right ventricle longitudinal strain | Baseline and 3-months (endpoint)
  Calculated from resting transthoracic echocardiographic (TTE) measurements using a portable ultrasound system (Siemens, USA) and a 4 mHz cardiac transducer. Reported as % or % per second.
Tricuspid annual plane systolic excursion (TAPSE) (mm) | Baseline and 3-months (endpoint)
  Calculated from resting transthoracic echocardiographic (TTE) measurements using a portable ultrasound system (Siemens, USA) and a 4 mHz cardiac transducer.
Fractional shortening (%) | Baseline and 3-months (endpoint)
  The reduction of the length of the end-diastolic diameter that occurs by the end of systole, calculated as: (((LVEDD - LVESD) / LVEDD)) * 100).

CONTACTS AND LOCATIONS:
Overall Officials: Craig Sale, PhD, Principal Investigator — Nottingham Trent University
Locations (2):
- United Kingdom (2):
  - Nottingham Trent University, Nottingham, Nottinghamshire
  - Aston University, Birmingham, West Midlands

IPD SHARING:
Plan to Share IPD: No
Research data will be deidentified and preserved for at least 10 years in an open-access data repository (e.g., Zenodo). This will allow anyone else (including other researchers and the general public) to also use the deidentified data for relevant analyses.